CLINICAL TRIAL: NCT01555437
Title: Assessment of Capsule Endoscopy Scoring Index, Clinical Disease Activity and Biological Markers in Small Bowel Crohn's Disease
Brief Title: Assessment of Capsule Endoscopy Scoring Index (CESI), Harvey-Bradshaw Index (HBI) and Biological Markers in Small Bowel Crohn's Disease (SBCD)
Status: Completed | Type: Observational
Sponsor: Shanghai Jiao Tong University School of Medicine (Other)
Responsible Party: Principal Investigator, Zhizheng Ge, Shanghai Institute of Digestive Disease，Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai Jiao Tong University School of Medicine
Other Study IDs: rjyyxhk0306
Record Dates: First submitted 2012-03-13; First posted 2012-03-15 (Estimated); Last update posted 2013-11-19 (Estimated); Status verified 2013-11

CONDITIONS: Small Bowel Crohn's Disease
Keywords: capsule endoscopy scoring index; Harvey-Bradshaw index; C-reactive protein; serum albumin; hemoglobin

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum of small bowel Crohn's disease patients
Oversight: Data Monitoring Committee: No

SUMMARY:
Background: Small bowel Crohn's disease (SBCD) is a chronic relapsing disease, and clinical presentation can vary considerably. Patients are frequently assessed by capsule endoscopy (CE), which enables direct visualization of small bowel mucosal abnormalities; however, the correlations between CE scoring index (CESI), biological markers, and disease activity indices remain undefined.

Methods: A prospective study was conducted between October 2008 and February 2011 on 58 established SBCD patients and suspected patients who received a definitive SBCD diagnosis during study. Patients underwent complete CE, and were scored according to the CESI (inactive, <135; mild inflammation, 135-790; moderate-severe inflammation, >790) and Harvey-Bradshaw index (HBI). Statistical correlation between CESI, HBI, C-reactive protein (CRP), serum albumin, and hemoglobin was assessed. At follow-up (~9 months), 11 of the patients underwent CE with scoring for CESI, HBI, and CRP.

DETAILED DESCRIPTION:
Parameters CESI To calculate the CESI, the small bowel was divided into three tertiles. The degree of disease involvement in each tertile was determined by assessing three parameters: villous edema, ulceration, and stenosis. Endoscopic remission was defined as CESI of <135. Mild inflammation was defined as CESI of 135-790, and moderate-severe inflammation as ≥790.

HBI HBI was used to assess the clinical disease activity. Patients with HBI >4 were considered to have clinically active disease.[7]

Blood analysis At the time of CE, patients provided a blood sample for measurement of hemoglobin, serum CRP, and albumin. Hemoglobin (normal ranges: women, 120-160 g/L and men, 140-180 g/L), albumin (normal range: 35-55 g/L), and CRP (upper limit of normal: <8 mg/L) were determined by routine laboratory tests.

ELIGIBILITY:
Inclusion Criteria:

* patients with known SBCD or newly diagnosed SBCD
* those patients for whom complete CE examination (in which the capsule
* reached the cecum within the CE test time) was achieved were retained for study

Exclusion Criteria:

* incomplete CE examination
* infectious enterocolitis
* symptoms related to perianal penetrating disease
* gastrointestinal cancer
* ulcerative colitis
* indeterminate colitis
* history of extensive small bowel resection
* known CD of the upper gastrointestinal tract or colon
* intake of non-steroidal anti-inflammatory drugs (NSAIDs) (more than two tablets per week)
* pregnancy

Ages: 17 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients underwent CE examination (described below), and only those patients for whom complete CE examination (in which the capsule reached the cecum within the CE test time) was achieved were retained for study.
Sampling Method: Probability Sample
Enrollment: 58 (Actual)
Dates: Start 2008-10; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Weak, but significant, correlations were found between CESI and HBI (r=0.4, p<0.01). | 2012.06
The correlation between CESI and CRP was moderate (r=0.58, p<0.01). | 2012.07
The median CRP value was significantly higher in patients with moderate-severe CESI, compared to the mild group (22.60±16.79 mg/L vs. 11.88±8.39 mg/L, p<0.01). | 2012.08
Changes between baseline and follow-up CESI failed to correlate with the delta-HBI or delta-CRP (both, p>0.05). | 2012.09

CONTACTS AND LOCATIONS:
Overall Officials: Zhizheng Ge, MD. Ph.D, Principal Investigator — RenJi Hospital